CLINICAL TRIAL: NCT07284420
Title: An ISA to Master Protocol ARGX-999-2-MG-2000 for an Exploratory, Phase 2a, Proof-of-Concept Study to Evaluate the Safety, Tolerability, and Efficacy of Empasiprubart IV as Add-On Therapy to Efgartigimod IV in Participants With AChR-Ab Seropositive Generalized Myasthenia Gravis With a Partial Clinical Response to Efgartigimod
Brief Title: ADAPT Forward 1 - ISA1 - a Study to Evaluate Empasiprubart IV as add-on Therapy to Efgartigimod IV in Participants With AChR-Ab Seropositive Generalized Myasthenia Gravis With a Partial Clinical Response to Efgartigimod
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-999-2-MG-20001; 2025-522492-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-08; First posted 2025-12-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: AChR-Ab Seropositive Generalized Myasthenia Gravis; Myasthenia Gravis; MG; gMG; Generalized Myasthenia Gravis; Generalized Myasthenia Gravis (gMG)
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod IV + Empasiprubart IV (Experimental): Participants receive efgartigimod IV in part A, B and C and empasiprubart IV in part B
  Interventions: Biological: Efgartigimod IV; Biological: Empasiprubart IV
- Efgartigimod IV (part A + C) (Experimental): Participants not eligible for part B, receiving efgartigimod IV in part A and C
  Interventions: Biological: Efgartigimod IV

INTERVENTIONS:
Biological: Efgartigimod IV — Intravenous infusion of efgartigimod
Biological: Empasiprubart IV — Intravenous infusion of empasiprubart
  Arms: Efgartigimod IV + Empasiprubart IV

SUMMARY:
This study is part of the ADAPT Forward platform study (NCT07294170). ADAPT Forward is a platform study with the aim to look at how safe different drugs are and how well they work for people with myasthenia gravis. The goal is to find the best therapeutic approach to reduce patients' side effects and improve their quality of life.

The aim of this ISA1 is to evaluate the safety and therapeutic relevance of empasiprubart as add-on therapy to efgartigimod in participants with AChR-Ab seropositive generalized myasthenia gravis.

The ADAPT Forward master protocol is registered on https://clinicaltrials.gov/study/NCT07294170

DETAILED DESCRIPTION:
Once the master protocol and ISA1 screening periods are completed, eligible participants can enroll in the run-in period (part A) where they will receive efgartigimod IV. Eligible participants can then continue to the add-on period (part B) where they will receive both efgartigimod IV and empasiprubart IV.

Participants who are not eligible for part B will continue directly to the safety follow-up period (part C) where they will receive efgartigimod IV only.

The study duration for each participant is approximately up to 54 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is seropositive for anti-acetylcholine receptor antibodies (AChR-Ab)
* Has confirmed diagnosis of gMG and is Myasthenia Gravis Foundation of America (MGFA) Class II, III, IVa, or IVb
* Has documented immunization against encapsulated bacterial pathogens (Neisseria meningitidis and Streptococcus pneumoniae) within 5 years of ISA screening or is willing to receive immunization at least 14 days before the first study drug administration

Exclusion Criteria:

* Clinical diagnosis of systemic lupus erythematosus (SLE)
* Any known complement deficiency
* Current administration of a complement inhibitor or received zilucoplan or eculizumab <2 months or ravulizumab <6 months before the first study drug administration
* Patients proven to be refractory to efgartigimod (ie, not achieving a clinically meaningful improvement in total Myasthenia Gravis Activities of Daily Living (MG-ADL) score defined as an improvement of ≥2 points)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2028-03-07 (Estimated); Study Completion 2028-03-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events in parts A and B | Up to 21 weeks

SECONDARY OUTCOMES:
MG-ADL total score change from baseline at week 18 in part B (cycle 2 day 29) compared with MG ADL total score change from baseline at week 4 in part A | Up to 18 weeks
  The Myasthenia Gravis Activities of Daily Living (MG- ADL) scale is an 8-item instrument used to assess MG symptoms and their effects on daily activities. The total score ranges from 0 (normal symptoms) to 24 (most severe symptoms)
Proportion of participants reaching MSE at any point in part B cycles 1 and 2, and part B cycles 1 or 2 | Up to 21 weeks
  MSE: Minimal symptom expression
MG-ADL total score changes from baseline over time in part B compared with part A | Up to 21 weeks
  The Myasthenia Gravis Activities of Daily Living (MG- ADL) scale is an 8-item instrument used to assess MG symptoms and their effects on daily activities. The total score ranges from 0 (normal symptoms) to 24 (most severe symptoms)
QMG total score change from baseline at week 18 in part B (cycle 2 day 29) compared with QMG total score change from baseline at week 4 in part A | Up to 18 weeks
  The Quantitative myasthenia gravis (QMG) includes 13 items that measure endurance or fatigability and accounts for fluctuations in disease state. The total score ranges from 0 (no disease severity) to 39 (highest disease severity)
QMG total score changes from baseline over time in part B compared with part A | Up to 21 weeks
  The Quantitative myasthenia gravis (QMG) includes 13 items that measure endurance or fatigability and accounts for fluctuations in disease state. The total score ranges from 0 (no disease severity) to 39 (highest disease severity)
Proportion of participants who have a 50% MG ADL total score improvement in part B cycles 1 and 2 | Up to 21 weeks
  The Myasthenia Gravis Activities of Daily Living (MG ADL) scale is an 8-item instrument used to assess MG symptoms and their effects on daily activities. The total score ranges from 0 (normal symptoms) to 24 (most severe symptoms)
Proportion of participants who have positive PASS in part B cycles 1 and 2, and part B cycles 1 or 2 | Up to 21 weeks
  PASS: Patient acceptable symptom state

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Profound Research LLC - Carlsbad, Carlsbad, California
  - Visionary Investigators Network, Miami, Florida
  - Dent Neurologic Institute - Amherst, Amherst, New York
  - Erlanger Health System, Chattanooga, Tennessee
  - National Neuromuscular Research Institute, Austin, Texas

IPD SHARING:
Plan to Share IPD: No